CLINICAL TRIAL: NCT01779596
Title: Effect of a Dual ET-blocker on Exercise Induced Blood Flow and Endothelial Function in T2DM
Brief Title: ET-blockade and Exercise Induced Blood Flow in T2DM
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Radboud University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: ET-EX-ACUTE
Record Dates: First submitted 2013-01-28; First posted 2013-01-30 (Estimated); Last update posted 2016-05-04 (Estimated); Status verified 2016-05

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: diabetes; endothelial function; exercise; blood flow; bosentan
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus; Motor Activity | interventions — Bosentan

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Bosentan (Experimental): Single dose of Bosentan (125 mg)
  Interventions: Drug: Bosentan
- Placebo (Placebo Comparator): Single dose of placebo (125 mg)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Bosentan
  Other Names: Tracleer; actelion pharmaceuticals; 125 mg oral dose
  Arms: Bosentan
Drug: Placebo
  Other Names: actelion pharmaceuticals; 125 mg oral dose
  Arms: Placebo

SUMMARY:
The purpose of this study is to establish the effect of ET blockade on the acute exercise induced blood flow and endothelial function in subjects with T2DM. We hypothesize that combining ET - blockade with exercise training leads to an acute increase of exercise induced blood flow when compared with exercise alone. We expect that this will lead to an optimization of vascular training effect in T2DM.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 Diabetes Mellitus (>2 years since diagnosis) OR controls

Exclusion Criteria:

* <40 years of age
* >65 years of age
* smoking
* cardiovascular disease
* diabetes related manifest vascular complications
* Type 1 Diabetes Mellitus
* use of Glibenclamide
* use of HIV drugs
* use of calcineurin inhibitors
* use of drugs that interfere with CYP3A4 and CYP2C19

Ages: 40 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2011-05; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
exercise induced blood flow | 2 hours

SECONDARY OUTCOMES:
exercise induced Flow Mediated Dilation | 2 hours

CONTACTS AND LOCATIONS:
Locations (1):
- Radboud University Nijmegen Medical Centre, Nijmegen, Gelderland, Netherlands

REFERENCES:
- [Derived] Schreuder TH, van Lotringen JH, Hopman MT, Thijssen DH. Impact of endothelin blockade on acute exercise-induced changes in blood flow and endothelial function in type 2 diabetes mellitus. Exp Physiol. 2014 Sep;99(9):1253-64. doi: 10.1113/expphysiol.2013.077297. Epub 2014 May 16. PMID 24928953